CLINICAL TRIAL: NCT05459129
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating The Efficacy and Safety of Multiple Treatment Combinations in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck (Morpheus-Head and Neck Cancer)
Brief Title: A Study Evaluating Efficacy and Safety of Multiple Treatment Combinations in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck (Morpheus-Head and Neck Cancer)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO43613
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — atezolizumab; Tiragolumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezo + Tira (Active Comparator): Participants in the atezolizumab plus tiragolumab arm will receive treatment for two cycles (6 weeks) until surgery or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Atezo + Tira + CP (Experimental): Participants in the atezolizumab plus tiragolumab plus carboplatin plus paclitaxel arm arm will receive treatment for two cycles (6 weeks) until surgery or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Tiragolumab — Tiragolumab will be administered intravenously at a fixed dose of 600 mg on Day 1 of each 21-day cycle.
Drug: Carboplatin — Carboplatin will be administered intravenously at a dose of area under the concentration-time curve (AUC) 5 mg/mL/min on Day 1 of each 21 day cycle.
  Arms: Atezo + Tira + CP
Drug: Paclitaxel — Paclitaxel will be administered intravenously at a dose of 175 mg/m2 on Day 1 of each 21 day cycle.
  Arms: Atezo + Tira + CP

SUMMARY:
This is a Phase Ib/II, open-label, multicenter, randomized, umbrella study in participants with locally advanced squamous cell carcinoma of the head and neck (SCCHN). The study will enroll treatment-naive participants with resectable Stage III-IVA human papillomavirus (HPV)-negative, programmed death-ligand 1 (PD-L1)-positive SCCHN with measurable disease, as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) who have not received systemic treatment for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Histologically confirmed, resectable Stage III-IVA SCCHN
* Eligible candidate for R0 resection with curative intent at the time of screening
* HPV-negative test for oropharyngeal carcinoma, as determined locally by p16 immunohistochemistry (IHC), in situ hybridization, or polymerase chain reaction-based assay
* Measurable disease (at least one target lesion), as assessed according to RECIST v1.1
* PD-L1 expression, defined as a combined positive score (CPS) >= 1
* Adequate hematologic and end-organ function
* Negative HIV test with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >= 200/μL, and have an undetectable viral load.
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following: Negative total hepatitis B core antibody (HBcAb), Positive total hepatitis B core antibody (HBcAb) followed by a negative quantitative hepatitis B virus (HBV) DNA.

Exclusion Criteria:

* HPV-positive oropharyngeal cancer, as determined locally by p16 IHC, in situ hybridization, or by polymerase chain reactions-based assay
* Distantly metastasized SCCHN
* Any prior therapy for SCCHN, including immunotherapy, chemotherapy, or RT
* Prior treatment with any of the protocol-specified study treatments
* Treatment with investigational therapy within 42 days prior to initiation of study treatment
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment or within 5 months after the final dose of study treatment
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT scan)
* History of malignancy other than SCCHN within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5 -year OS rate>90%)
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic or prophylactic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment
* Significant cardiovascular disease such a New York Heart Association cardiac disease (Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhytmia, or unstable angina
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to study initiation of study treatment, or anticipation of need for a major surgical procedure other than tumor resection, during the study
* Any of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of investigational drug, may affect the interpretation of the results, impair the ability of the patient to participate in the study, or renders the patient at high risk form treatment complications
* History of severe allergic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies
* Known allergy or hypersensitivity to any of the study drugs or their excipients
* Known intolerance to any of the drugs required for premedication
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Eligible only for the control arm
* Active EBV infection or known or suspected chronic EBV infection at screening

Specific Exclusion Criteria for Atezo+Tira+CP:

* Known severe allergy or hypersensitivity to placlitaxel, platinum or platinum-containing compounds
* Known history of severe hypersensitivity to products containing Cremophor EL
* Creatinine clearance <45m./min (Calculated using the Cockcroft-Gault formula)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (3):
  - City of Hope, Duarte, California
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Hadassah University Hospital - Ein Kerem, Jerusaelm, Israel
- South Korea (2):
  - Severance Hospital - Yonsei Cancer Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants with locally advanced squamous cell carcinoma of the head and neck (SCCHN) took part in the study across 6 investigative sites in Israel, the Republic of Korea, and the United States from 12 April 2023 to 15 Aug 2024.
Pre-assignment Details: Participants were randomized to receive either Atezolizumab + Tiragolumab or Atezolizumab + Tiragolumab + carboplatin/ paclitaxel (CP). At the discretion of the investigator, participants started adjuvant therapy outside of this study, commencing between Week 10 and Week 13 and after treatment completion/discontinuation visit.
Groups:
- Atezolizumab + Tiragolumab: Participants received atezolizumab, 1200 milligrams (mg) as intravenous (IV) infusion, along with tiragolumab, 600 mg, as IV infusion on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7 ± 1 week) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
- Atezolizumab + Tiragolumab + CP: Participants received atezolizumab, 1200 mg as IV infusion, along with tiragolumab, 600 mg, as IV infusion; carboplatin, at a dose of AUC 5 mg/mL/min as IV infusion and paclitaxel, 175 mg/m^2, as IV infusion on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7 ± 1 week) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
Period: Overall Study
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Death | 1 | 0
Not completed — Study Terminated By Sponsor | 5 | 6

BASELINE CHARACTERISTICS:
Population: Safety-evaluable population included all randomized participants who received any amount of dose of any component of the study treatment.
Groups:
- Atezolizumab + Tiragolumab: Participants received atezolizumab, 1200 mg as IV infusion, along with tiragolumab, 600 mg, as IV infusion on Day 1 of each 21-day cycle for 2 cycles (6 weeks) until surgery (Week 7 ± 1 week) or until unacceptable toxicity or loss of clinical benefit, whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.83 (8.68) | 52.33 (9.65) | 60.08 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathologic Complete Response (pCR) as Determined by Local Pathologic Review
Description: pCR was defined as the absence of any viable primary tumor at time of surgical resection, as determined by local pathologic review. The pCR rate was defined as the percentage of participants who achieved a pCR. pCR rate was calculated for each arm, along with the 95% confidence interval (CI) estimated using the Clopper-Pearson method and the 95% CI for difference in rates was estimated using the Wald method with continuity correction. Participants with missing or no pathologic response assessment were classified as non-responders. Percentages have been rounded off to the nearest whole number.
Time Frame: At the time of surgery (Week 7 ± 1 week)
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
percentage of participants | 16.7 [0.42 to 64.12] | 50.0 [11.81 to 88.19]
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; Test type: Superiority; Difference in pCR Rates = 33.33, 95% CI 2-sided [-33.23 to 99.90]

2. Secondary Outcome: Pathologic Response Rate (pRR) as Determined by Local Pathologic Review
Description: pRR was defined as the percentage of participants with a pCR, major pathological response (mPR), and pathological partial response (pPR). pCR was defined as the absence of any viable primary tumor at time of surgical resection, as determined by local pathologic review. mPR was defined as ≤10% residual viable tumor at the time of surgical resection in the primary tumor. pPR was defined as ≤ 50% residual viable tumor at the time of surgical resection in the primary tumor. pRR was calculated for each arm, along with the 95% CI, estimated using the Clopper-Pearson method, and the 95% CI for the difference in rates was estimated using the Wald method with continuity correction. Percentages have been rounded off to the nearest whole number.
Time Frame: At the time of surgery (Week 7 ± 1 week)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
percentage of participants | 66.7 [22.28 to 95.67] | 100 [54.07 to 100.00]
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; Test type: Superiority; Difference in pRR = 33.33, 95% CI 2-sided [-21.05 to 87.72]

3. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from randomization to disease progression (PD) that precludes surgery, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1); local, regional, or distant disease recurrence or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), and must also demonstrate an absolute increase of ≥ 5 millimeters (mm). Kaplan-Meier method was used to estimate the median for EFS, and 95% Cls was constructed using Brookmeyer and Crowley method. Data from participants who have not experienced such events were censored at the time of the last tumor assessment. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made in terms of median EFS per arm or HR between the arms.
Time Frame: From randomization to PD disease recurrence or death (Up to 9.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
months | NA [2.96 to NA] — Median and upper and lower limits of 95% CI could not be estimated due to insufficient events as the study was terminated prematurely | NA [4.30 to NA] — Median and upper and lower limits of 95% CI could not be estimated due to insufficient events as the study was terminated prematurely
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; Test type: Superiority; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.11 to 3.91] — HR was estimated by Cox regression. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made in terms of median EFS per arm or HR between the arms

4. Secondary Outcome: Relapse-Free Survival (RFS)
Description: RFS was defined as the time from surgery to the first documented recurrence of disease or death from any cause. Recurrent disease included local, regional, or distant recurrence: local recurrence was defined as tumor regrowth within 2 centimeter (cm) of the primary lesion's tumor bed; regional recurrence as any nodal or non-nodal tumor lesions that are more than 2 cm from the primary lesion but are not beyond the regional nodal basin; distant recurrence as any non-local/non-regional recurrence. Participants who did not have documented recurrence of disease or died, RFS was censored at the day of the last tumor assessment. Kaplan-Meier method was used to estimate the median for RFS, and 95% Cls was constructed using Brookmeyer and Crowley method. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made in terms of median RFS per arm or HR between the arms.
Time Frame: From surgery (scheduled at Week 7 ± 1 week) to first documented disease recurrence or death (up to 7.6 months)
Population: Adjuvant-evaluable population included all participants who received at least one dose of each drug and who completed surgery.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 5 | 6
months | NA [0.99 to NA] — Median and upper limit of 95 % CI was not estimable due to insufficient number of participants with events. | NA [2.79 to NA] — Median and upper limit of 95 % CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.13 to 6.43] — HR was estimated by Cox regression. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made in terms of media RFS per arm or HR between the arms

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause. Data from participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. Kaplan-Meier method was used to estimate the median for OS, and 95% Cls was constructed using Brookmeyer and Crowley method. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made in terms of median OS and no further OS analysis are reported.
Time Frame: From randomization to death from any cause or last known to be alive (Up to 9.2 months)
Population: Efficacy-evaluable population included all who received at least one dose of each drug for their assigned treatment regimen.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
months | NA [NA to NA] — Median and 95 % CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — Median and 95 % CI was not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with an objective tumor response of complete response (CR) or partial response (PR) as determined by the investigator using RECIST v.1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. ORR was calculated for each arm, along with 95% CIs, using the Clopper-Pearson method and the 95% CI for difference in rates was estimated using the Wald method with continuity correction. Participants with missing or no response assessments were classified as non-responders.
Time Frame: Prior to surgery (up to Week 6)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
percentage of participants | 33.3 [4.33 to 77.72] | 50.0 [11.81 to 88.19]
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; Test type: Superiority; Difference in ORR = 16.67, 95% CI 2-sided [-54.99 to 88.32]

7. Secondary Outcome: Landmark EFS Rate
Description: EFS was defined as the time from randomization to PD that precludes surgery, as determined by the investigator according to RECIST v1.1; local, regional, or distant disease recurrence or death from any cause, whichever occurs first. EFS rate was defined as the percentage of participants who are event-free at the specified timepoints. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline), and must also demonstrate an absolute increase of ≥ 5 mm. Landmark EFS rates were estimated for each study arm using the Kaplan-Meier method, with 95% CIs calculated through the use of Greenwood's formula. Percentages have been rounded off to the nearest whole number. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made.
Time Frame: 3 Months, 6 Months, and 1 Year
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an EFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
percentage of participants
  3 Months: number analyzed (Participants) | 4 | 5
  3 Months | 66.67 [28.95 to 100.00] | 83.33 [53.51 to 100.00]
  6 Months: number analyzed (Participants) | 4 | 4
  6 Months | 66.67 [28.95 to 100.00] | 66.67 [28.95 to 100.00]
  1 Year: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; 3 Months Analysis; Test type: Superiority; Difference in Event Free Rate = 16.67, 95% CI 2-sided [-31.42 to 64.75] — Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made
Statistical Analysis 2: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; 6 Months Analysis; Test type: Superiority; Difference in Event Free Rate = 0.00, 95% CI 2-sided [-53.34 to 53.34] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Landmark RFS Rate
Description: RFS was defined as the time from surgery to the first documented recurrence of disease or death from any cause. RFS rate was defined as the percentage of participants who are event-free at the specified timepoints. Recurrent disease included local, regional, or distant recurrence: local recurrence was defined as tumor regrowth within 2 cm of the primary lesion's tumor bed; regional recurrence as any nodal or non-nodal tumor lesions that are more than 2 cm from the primary lesion but are not beyond the regional nodal basin; distant recurrence as any non-local/non-regional recurrence. Landmark RFS rates were estimated for each study arm using the Kaplan-Meier method, with 95% CIs calculated through the use of Greenwood's formula. Percentages have been rounded off to the nearest whole number. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made .
Time Frame: 3 Months, 6 Months, and 1 Year
Population: Adjuvant-evaluable population included all participants who received at least one dose of each drug and who completed surgery. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an RFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 5 | 6
percentage of participants
  3 Months: number analyzed (Participants) | 4 | 4
  3 Months | 80.00 [44.94 to 100.00] | 66.67 [28.95 to 100.00]
  6 Months: number analyzed (Participants) | 2 | 2
  6 Months | 60.00 [17.06 to 100.00] | 66.67 [28.95 to 100.00]
  1 Year: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; 3 Months Analysis; Test type: Superiority; Difference in Event Free Rate = -13.33, 95% CI 2-sided [-64.83 to 38.16] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Atezolizumab + Tiragolumab vs Atezolizumab + Tiragolumab + CP; 6 Months Analysis; Test type: Superiority; Difference in Event Free Rate = 6.67, 95% CI 2-sided [-50.49 to 63.82] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Landmark OS Rate
Description: OS was defined as the time from randomization to death from any cause. OS rate was defined as the percentage of participants who are event-free at the specified timepoints. Landmark OS rates were estimated for each study arm using the Kaplan-Meier method, with 95% CIs calculated through the use of Greenwood's formula. Due to the early termination of the study, the limited sample size and follow-up time no meaningful conclusions can be made .
Time Frame: 3 Months, 6 Months, and 1 Year
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an OS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
percentage of participants
  3 Months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  6 Months: number analyzed (Participants) | 5 | 6
  6 Months | 83.33 [53.51 to 100.00] | 100.00 [100.00 to 100.00]
  1 Year: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: From initiation of study treatment up to 135 days after the final dose of study treatment (up to 5.1 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

11. Secondary Outcome: Number of Participants With Immune-Related AEs Grade >=3
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Grade 3 AEs were defined as severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living.
Time Frame: Up to 12 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

12. Secondary Outcome: Rate of Delayed Surgery Due to Treatment-Related AEs
Description: Rate of delayed surgery due to treatment related AEs was defined as the percentage of participants for whom surgery was delayed due to treatment-related AEs for 2 weeks. An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Delay up to week after the planned time of surgery (scheduled at Week 7 ± 1 week) up to 2 weeks (up to Week 9)
Population: Safety-evaluable population included all randomized participants who received any amount of dose of any component of the study treatment. Percentages have been rounded off.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

13. Secondary Outcome: Duration of Delayed Surgery Due to Treatment-Related AEs
Description: Duration of surgery delay due to treatment related AEs was calculated on the participants for whom surgery was delayed due to treatment-related AEs for 2 weeks. An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Delay up to week after the planned time of surgery (scheduled at Week 7 ± 1 week) up to 2 weeks (up to Week 9)
Population: Safety-evaluable population included all randomized participants who received any amount of dose of any component of the study treatment. No participants had surgery delayed due to treatment-related AEs.
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Rate of Surgical Complications as Assessed According to the Clavien-Dindo Surgical Classification
Description: Surgical complications were scored according to Clavien-Dindo surgical classification. Complication rates for every grade were reported & scored for participants who underwent complete lymph node dissection (CLND). The Surgical complications according to Clavien-Dindo can be classified into following grades: Grade I: Any complication that does not need pharmacological treatment or surgical, endoscopic, and radiological interventions. Grade II: Complications that require pharmacological treatment with drugs or blood transfusions and total parenteral nutrition. Grade III: Complications that require surgical, endoscopic, or radiological intervention with (Grade IIIb) or without (Grade IIIa) general anesthesia. Grade IV: Life-threatening complications requiring intensive care unit (ICU) management, which may be single organ (Grade IVa) or multiorgan (Grade IVb) dysfunction. Grade V: Complications that might cause the death of a participant. Only categories with non-zero data was reported.
Time Frame: From Surgery (Week 7 ± 1 week) up to 5.1 months
Population: Safety-evaluable population included all randomized participants who received any amount of dose of any component of the study treatment. Overall number analyzed is the number of participants who underwent surgery. Percentages have been rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
Number analyzed (Participants) | 5 | 6
percentage of participants | 0 | 16.7

ADVERSE EVENTS:
Time Frame: From initiation of study treatment up to 135 after the final dose of study treatment (up to 5.1 months) All-cause mortality: Up to 9.2 months
Description: Safety-evaluable population included all randomized participants who received any amount of dose of any component of the study treatment.
Arm/Group | Atezolizumab + Tiragolumab | Atezolizumab + Tiragolumab + CP
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Tiragolumab (N=6) | Atezolizumab + Tiragolumab + CP (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vascular rupture (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Tiragolumab (N=6) | Atezolizumab + Tiragolumab + CP (N=6)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (7)
Oral pain (Gastrointestinal disorders) | 1 (2) | 3 (3)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 2 (4)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT05459129/Prot_SAP_000.pdf